CLINICAL TRIAL: NCT04610437
Title: Fixation of Digital Arthrodesis With Percutaneous Kirschner Wire Versus Intramedullary Fixation With Resorbable Polylactic Acid Needle: A Comparative Study
Brief Title: Intramedullary Resorbable Fixation System Versus K-wire for the Treatment of Lesser Toe Deformities
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Seville (Other)
Responsible Party: Principal Investigator, Manuel Coheña-Jiménez, PhD- principal investigator and clinical professor, University of Seville
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: University of Seville-USeville
Record Dates: First submitted 2020-10-22; First posted 2020-10-30 (Actual); Last update posted 2020-11-17 (Actual); Status verified 2020-11

CONDITIONS: Hammer Toe; Surgery; Deformity of Toe; Phalanx; Dislocation Toe(S)
Keywords: arthodesis; kirschner wire; PLLA
MeSH Terms: conditions — Hammer Toe Syndrome

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intramedullary reabsorbable fixation system PLLA. (Active Comparator): Arthrodesis interphalangeal with intramedullary reabsorbable fixation system PLLA.
  Interventions: Procedure: Arthrodesis interphalangeal with intramedullary resorbable fixation system
- K-wire (Placebo Comparator): Arthrodesis interphalangeal with kirschner wire
  Interventions: Procedure: Arthrodesis interphalangeal with intramedullary resorbable fixation system

INTERVENTIONS:
Procedure: Arthrodesis interphalangeal with intramedullary resorbable fixation system — Interphalangeal arthrodesis of lesser toes with two different fixation systems.
  Other Names: Arthrodesis interphalangeal with kirschner wire fixation system

SUMMARY:
Hammertoe deformity is one of the most common deformities in the foot and is characterized by dorsiflexion of the proximal phalanx at the metatarsal-phalangeal joint and a plantarflexion of the middle phalanx at the proximal interphalangeal joint. Surgical intervention for this type of deformity is indicated when the symptoms progress and conservative treatments are not enough, that is, when we are faced with a rigid painful deformity.Arthrodesis of the proximal interphalangeal joint temporarily fixed with a Kirschner wire is the most commonly used techniques.

Therefore, intramedullary fixation with a PLLA needle may be a good alternative. The use of biomaterial is gaining relevance in foot surgery, with polylactic acid being the most widely used due to its strength. Its total biodegradation requires a time of 16-24 months. No cases of foreign body reaction have been described with this type of osteosynthesis material, due to its characteristics similar to those of bone. Its only drawbacks are that it increases the complexity of the technique and that it increases the cost of the procedure. Being a flexible needle, it allows to leave a functional intraoperative claw. It maintains the functionality of the distal interphalangeal joint and carries a lower risk of infection by carrying osteosynthesis material on the outside.

The purpose of the present study is to prospectively collect clinical and radiographic outcomes of operative correction of hammertoe deformity using a fixation system of intramedullary device of polylactic acid versus a kirschner wire.

DETAILED DESCRIPTION:
A comparative, prospective, randomised study.

ELIGIBILITY:
Inclusion Criteria:

* Clinical and radiological evidence of rigid hammer toe.
* Non-smoking patient.
* Have no previous surgical episode or known trauma to the foot or ankle of the same limb.
* Not have any significant medical comorbidity:
* Uncontrolled hypertension.
* Previous myocardial infarction.
* Neoplasms.
* Chronic obstructive pulmonary disease.
* Arrhythmias.
* Morbid obesity.
* Uncontrolled diabetes mellitus.
* Peripheral vascular disease.
* Peripheral neuropathy.
* Lumbar disc herniation.
* Any neuro-muscular alteration.
* That the patient present:
* Palpable peripheral pulses through the posterior tibial artery and pedia.
* Ankle-brachial index or YAO between 1-1.2.
* Partial oxygen saturation> or = 95%.

Exclusion Criteria:

* That the patient has undergone another previous surgical procedure on the same foot.
* Known trauma to the foot to be intervened.
* History of sensitivity to local anesthetics.
* Pregnant or lactating women.
* Follow-up time less than 90 days.
* Patients with any systemic pathology or in chronic treatment that could interfere with the favorable evolution of the process.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2019-05-23 (Actual); Study Completion 2020-09-30 (Actual)

PRIMARY OUTCOMES:
Change of AOFAS MTP-IP for the lesser toes | baseline, 6 weeks, 6 months
  Each measure is comprised of nine questions and cover three categories: Pain (40 points), function (50 points) and alignment (10 points). These are all scored together for a total of 100 points.

SECONDARY OUTCOMES:
Change of Finger alignment. | Baseline, 6 weeks, 6 months
  X-ray in dorsal-plantar projection in load to measure the angle formed between the longitudinal axes of the proximal and middle phalanges. Good: 0-10º. (tb smartoe vs kw buried and the other from smartoe); Enough: 11-20º; or Bad:> 20º.
Change of visual analog scale | Baseline, 6 weeks, 6 months
  Heel pain intensity was referred to as 0-10, in which 0= no pain at all and 10= the worst pain possible
Level of Satisfaction | Baseline, 6 weeks, 6 months
  Satisfaction assessed by the scale.This is a self-administered scale of satisfaction with the procedure with 4 categories. The response categories consisting of very satisfied (4 points), somewhat satisfied (3 points), somewhat dissatisfied ( 2 points), and very dissatisfied (1 points).
Change of Foot health status questionnaire | Baseline, 6 weeks, 6 months
  Foot Health Status Questionnaire: The questionnaire to measure foot health related quality of life. The Foot Health Status Questionnaire Data Analysis Software obtain the scale scores for the domains of; Foot Pain, Foot Function, Footwear, General Foot Health Perceptions from respondent's answers on the questionnaire.The questionnaire does not providean overall score. To obtain these indexes, the responsesare analysed through computer software (FHSQ, version1.03). After processing the data, the software produces ascore ranging from 0 to 100. The maximum score is in-dicative of a person with excellent foot health, no painor discomfort and no difficulty or limitations in puttingon shoes, performing activities of daily life or work, with adequate functional capacity; a score of zero representsthe worst state of health for the foot.

CONTACTS AND LOCATIONS:
Overall Officials: Pedro Montaño Jiménez, PhD, Study Director — University of Seville; Luis María Gordillo Fernández, PhD, Study Director — University of Seville; Juan Manuel Muriel Sánchez, Principal Investigator — University of Seville; Manuel Coheña Jiménez, PhD, Study Director — University of Seville
Locations (1):
- Manuel Coheña Jiménez, Seville, Spain

IPD SHARING:
Plan to Share IPD: No